CLINICAL TRIAL: NCT01608412
Title: An Open-label Randomized Controlled Clinical Trial to Assess the Efficacy and Safety of the Conversion to Everolimus 3 Months After Kidney Transplantation.
Brief Title: A Clinical Trial to Assess the Efficacy and Safety of the Conversion to Everolimus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001ABR19T
Record Dates: First submitted 2012-05-08; First posted 2012-05-31 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2011-08

CONDITIONS: Kidney Transplant Recipients
Keywords: renal transplantation; everolimus; tacrolimus; molecular evaluation
MeSH Terms: interventions — Tacrolimus; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus (Active Comparator): The subjects included in the study will be clinically followed up for at least 12 months. The patients will be selected at 3 months post-transplant according to inclusion and exclusion criteria and randomized in a 1:1 ratio for conversion to everolimus or maintenance of tacrolimus therapy.
  Intervention arm: Tacrolimus
  Interventions: Drug: Tacrolimus
- Everolimus (Active Comparator): The subjects included in the study will be clinically followed up for at least 12 months. The patients will be selected at 3 months post-transplant according to inclusion and exclusion criteria and randomized in a 1:1 ratio for conversion to everolimus or maintenance of tacrolimus therapy.
  Intervention arm: Everolimus
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Tacrolimus — TACROLIMUS (C0 = 5-10 ng/mL) + MPS 1440 mg + Pred
  Arms: Tacrolimus
Drug: Everolimus — Everolimus (C0 = 6-10 ng/mL) + MPS 1440 mg + Pred
  Arms: Everolimus

SUMMARY:
The study hypotheses to be tested in this study are:

* Conversion to everolimus at 3 months post-transplantation is safe and effective;
* Accurate noninvasive molecular diagnostic tests can replace biopsy at 3 months pre-conversion (for the diagnosis of subclinical cellular and/or humoral rejection, tissue fibrosis and calcineurin inhibitor-induced nephrotoxicity) in kidney transplant recipients;
* Follow-up biopsy at 12 months post-conversion (for the diagnosis of tissue fibrosis) can be replaced with accurate noninvasive molecular diagnostic tests in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing their first living- or deceased-donor kidney transplant who maintain a functioning graft 3 months post-transplant;
* Older than 18 years;
* Panel-reactive antibodies lower than 20%;
* Baseline immunosuppression with tacrolimus, mycophenolate sodium (MPS) and prednisone at randomization at 3 months.

Exclusion Criteria:

* eGFR < 35 mL/min at randomization;
* Urine protein-to-creatinine ratio > 0.8 at randomization;
* Episode of acute rejection with Banff histological classification > 1A in the first 3 months post-transplant;
* Cholesterol > 350 mg/dL or triglycerides > 400 mg/dL with therapy at randomization;
* Active infection at randomization;
* Chronic liver disease;
* Refusal to participate in the study;
* Contraindications to kidney biopsy;
* Biopsy findings at 3 months post-transplant including borderline rejection, cellular rejection or antibody-mediated rejection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate cumulative patient and graft survival at 12 months post conversion | one year
  Patient and graft survival will be evaluated one year after randomization by Kaplan-Meier analysis

SECONDARY OUTCOMES:
Evaluation of estimated glomerular filtration rate 12 months post-conversion | one year
  - To assess the efficacy of conversion from tacrolimus to everolimus 12 months post-conversion by measuring the estimated glomerular filtration rate using the Modification of Diet in Renal Disease (MDRD) equation

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Felipe S. Gonçalves, MD, Principal Investigator — HCPA
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil